CLINICAL TRIAL: NCT05948371
Title: Effects of High Intensity Aerobic Interval Training Versus Continuous Training in Heart Failure Patients.
Brief Title: High Intensity Aerobic Interval Training Versus Continuous Training in Heart Failure Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/01653 Hafiza Misbah Inayat
Record Dates: First submitted 2023-07-07; First posted 2023-07-17 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Intensity interval Training (Experimental)
  Interventions: Other: High Intensity interval Training
- Continuous Aerobic training (Active Comparator)
  Interventions: Other: Continuous Aerobic training

INTERVENTIONS:
Other: High Intensity interval Training — High Intensity interval Training
  * Frequency: 3-5 day per week
  * Intensity: 60 to 80% of HRR. If atrial fibrillation present use RPE of 11-14 on a 6-20 scale.
  * Time: total 30 mint time.6 mint exercise with high intensity and 2 mints of low intensity for active recovery until 30 mints complete.
  Type: walking and static cycling. Walking
  * Frequency 3 -5 days per week Intensity : use RPE of 11-14.
  * Time:30 mint total. 6 mint walk with high intensity and 2 mint walk with low intensity until 30mints completed.
  Arms: High Intensity interval Training
Other: Continuous Aerobic training — Continuous Aerobic training
  * Frequency : 3-5 days per week.
  * Intensity:40-70% of HHR.
  * Time : initial 5-10 then 10-15 until 30mints without rest interval
  * Type : walking and static cycling.
  Arms: Continuous Aerobic training

SUMMARY:
To determine the effect of high intensity aerobic interval training versus continuous aerobic training in heart failure patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient with heart failure including both male and female
* Patients who can perform 6 MWT.
* According to classification of American heart association, class 1 heart failure patients are included.

Exclusion Criteria:

* Heart failure patients along with orthopedic problems.
* Patients who have use pacemaker.
* Patient who have recent acute myocardial infraction or revascularization less than 3 months.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
6MWT Distance | 8 week
  Changes from the baseline, 6 min walk test was used to measure Functional capacity. It is a sub maximal exercise test which can aid in assessing functional capacity of patients with cardiopulmonary diseases, in this test we find out the maximum distance in meters which an individual covers in 6 min.
Minnesota living with heart failure questionnaire | 8 week
  MLWHFQ is commonly used health related quality of life questionnaires with heart failure. This is very easy to apply on patients and self-administered questionnaire. It has two components emotional and physical and total score. Each item is scored in a 6.likert scale (0 to 5), thus, the total score could range from 5 to 105, with higher scores indicating more significant impairment in health related quality of life. Changes from the basline will be measured
Pulse Rate | 8 week
  Changes from baseline, Pulse rate was measured per minute through pulse oximeter
Oxygen Saturation (SpO2) | 8 week
  Changes from baseline SPO2 was measured in percentage. Oxygen immersion is the division of oxygen-soaked hemoglobin with respect to add up to hemoglobin in the blood. Pulse oximeter measure it.
Modified Borg dyspnea scale | 8 week
  Changes from the Baseline, It is a subjective numeric scale ranging from 0 to 10, where 0 indicates "no dyspnea" and 10 indicates "unbearable dyspnea." A number is chosen by the patient in order to decide the best score that matches his level of dyspnea during physical activity.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Iqbal Tariq, PhD*, Principal Investigator — Riphah International University
Locations (1):
- Railway General Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No